CLINICAL TRIAL: NCT06182293
Title: Impact of Systemic Sclerosis on the Periodontal Microbiota: a Pilot Study
Brief Title: Periodontal Microbiota in Systemic Sclerosis
Acronym: Periomicross
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9149
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Scleroderma Systemic
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic sclerosis (Other)
  Interventions: Other: Subgingival dental plaque sampling for whole metagenome sequencing of the periodontal microbiota
- Controls (Other)
  Interventions: Other: Subgingival dental plaque sampling for whole metagenome sequencing of the periodontal microbiota

INTERVENTIONS:
Other: Subgingival dental plaque sampling for whole metagenome sequencing of the periodontal microbiota — Subgingival plaque will be collected at 6 sites using sterile curettes after removal of supragingival biofilm by brushing. After microbial DNA extraction, whole metagenome will be sequenced.

SUMMARY:
Systemic sclerosis (SSc) is a rare and complex autoimmune disease. Although its etiology remains unknown, various environmental factors, including certain microorganisms, can represent potential triggers of SSc in individuals with a permissive genetic background. Patients show a wide spectrum of clinical features including periodontitis, which is an inflammatory disease of the tooth-supporting tissues resulting from dysbiosis of the periodontal microbiota guided by inflammophilic bacteria.

The microbiota plays a fundamental role in the induction, training, and function of the host immune system. Numerous studies have highlighted the impact of an altered microbiota, i.e. dysbiosis, on the pathogenesis of immune-mediated diseases. Indeed, commensals are important to maintain immune homeostasis and changes in the microbial composition can be responsible for a loss of tolerance. SSc has been shown to be associated with gut dysbiosis and a depletion of commensals. However, although the oral cavity is one of the two largest microbial habitats, only one study (only focusing on Lactobacillus species) has investigated the oral microbiota in SSc. As periodontal dysbiosis is known to induce low-grade systemic inflammation and represents a risk factor for the development of various autoimmune diseases, the relationship between periodontal microbiota composition and SSc merits further exploration.

The aim of this pilot study is to characterize the taxonomic composition and metabolic pathways of the periodontal microbiota in SSc patients and age and sex-matched controls.

ELIGIBILITY:
Inclusion Criteria:

Common inclusion criteria

* Men or women over 18 (adults)
* Affiliation to a social health insurance plan
* Subject able to understand the aims and risks of the research and to give signed informed consent form prior to the inclusion in the study
* More than 12 teeth suitable for evaluation

Inclusion criteria for systemic sclerosis patients

* Systemic sclerosis patient with a diagnosis based on the American College of Rheumatology/European League Against Rheumatism criteria (LeRoy et al., 1988 ; van den Hoogen et al., 2013)
* Diagnosis made during the 2 years preceding study inclusion (early form of the disease)

Inclusion criteria for controls

- Patient attending the Oral Medicine and Surgery Department from the University Hospital of Strasbourg for a routine dental consultation

Exclusion Criteria:

* - Subject under court protection
* Subject under guardianship or curatorship
* Pregnancy or breastfeeding
* Impossibility to provide accurate information (emergency situation, comprehension difficulties…)
* Subject currently involved in another clinical trial or in an exclusion period following participation in another clinical trial
* Smoking (≥ 10 cigarettes per day)
* Other associated systemic auto-immune disease (Sjögren syndrome with positive serum anti-SSA and/or anti-SSB auto-antibodies, systemic lupus erythematosus…)
* Progressive chronic illness other than systemic sclerosis
* Acute infection at inclusion
* Progressive cancer or cancer diagnosed within 2 years prior to the study
* Ongoing antibiotic and/or antifungal treatment or within 3 months prior to inclusion
* Probiotics and/or prebiotics intake within 3 months prior to inclusion
* Oral antiseptics within the week before inclusion (chlorhexidin mouthwashes…)
* Risk of infective endocarditis
* Corticosteroids ≥10 mg/day and/or proton pump inhibitors within 3 months prior to inclusion
* Previous hematopoietic stem cell transplantation
* Another cause of skin sclerosis (radiotherapy of the orofacial area…)
* Periodontal specialized treatments, root and/or periodontal surgical treatment and/or subgingival instrumentation within the year before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity of the periodontal microbiota using Chao-1 index | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Dentaire, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No